CLINICAL TRIAL: NCT03144960
Title: Mechanical Thrombectomy Of Acute Occlusion In Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHMohamed, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thrombectomy
Record Dates: First submitted 2017-04-17; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mechanical thrombectomy (Other): The study will be performed involving ischemic stroke patients with proximal occlusion within 4.5 hours from stroke onset, mechanical thrombectomy with retrievable stents, thrombus aspiration, retraction, wire disruption.
  Interventions: Procedure: Mechanical Thrombectomy

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — mechanical thrombectomy with retrievable stents, thrombus aspiration, retraction, wire disruption

SUMMARY:
Assessment of Therapeutic benefits and hazards of Mechanical Thrombectomy in Ischemic stroke patients with proximal occlusion within 4.5 hours from stroke onset.

DETAILED DESCRIPTION:
Stroke is an acute neurologic dysfunction of vascular origin with sudden or at least rapid occurrence of symptoms and signs corresponding to the involvement of focal areas in the brain.The two main types of stroke are ischemic and hemorrhagic.Thrombosis can form in the extracranial and intracranial arteries when the intima is roughened and plaque forms along the injured vessel.The endothelial injury permits platelets to adhere and aggregate, then coagulation is activated and thrombus develops at site of plaque.Blood flow through the extracranial and intracranial systems decreases, and the collateral circulation maintains function. When the compensatory mechanism of collateral circulation fails, perfusion is compromised, leading to decreased perfusion and cell death. Stroke is the third leading cause of death in the United States. Many people die each year from stroke in the United States.Stroke is the leading cause of serious, long-term disability in the United States. Nearly one fourth of strokes occur in people under the age of 65.High blood pressure is the most important risk factor for stroke. Intravenous recombinant tissue-type plasminogen activator is the only Food and Drug Administration approved treatment for acute ischemic stroke. Mechanical thrombectomy improves clinical outcomes in patients with acute ischemic stroke caused by a large vessel occlusion.There is no apparent benefit of intravenous thrombolysis to patients with ischemic stroke undergoing mechanical thrombectomy. The study will be performed involving ischemic stroke patients with proximal occlusion within 4.5 hours from stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 - 80 years old of both sex.
2. Acute ischemic stroke due to proved large-artery occlusion.
3. Ineligibility for IV thrombolysis.
4. A timeframe of ≤ 4.5 hours between stroke onset and the start of mechanical thrombectomy.
5. The patients included in this series should have an NIHSS score of at least 10 or fluctuating symptoms.
6. ASPECTS of 6 or > 6
7. All patients will be undergoing CT/CT angiography before and after treatment

Exclusion Criteria:

1. Age older than 80 years or less than 18
2. Cerebral haemorrhage.
3. Acute infarction > 1/3 of middle cerebral artery (MCA) territory on CT-scan.
4. A history of stroke in the last 6 weeks.
5. A time interval of > 4.5 hours.
6. laboratory evidence of coagulation abnormalities.
7. Known arteriovenous malformation , neoplasm or aneurysm.
8. Woman at child bearing age who has a positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Of Acute Occlusion In Ischemic Stroke by Mechanical Thrombectomy | 18 months
  Treatment of ischemic stroke patients after 4.5 hours from stroke onset by endovascular intervention by using Mechanical Thrombectomy techniques and without using Recombinant tissue-type plasminogen Activator and non eligible patients for Thrombectomy will be excluded.
  The number of people will be participated into this study will be 20 aged 18 to 80 years old The patients will be undergoing NIHSS score , ASPECTS score The patients will be undergoing CT/CT angiography The patients will be undergoing mechanical thrombectomy Results will be collected and correlated with the prognosis of the outcomes

SECONDARY OUTCOMES:
The patients will be undergoing NIHSS score | 1 hour
  patients with NIHSS score less than 10 non eligible for mechanical thrombectomy
The patients will be undergoing ASPECTS score | 1 hour
  patients with ASPECTS score less than 6 non eligible for mechanical thrombectomy
The patients will be undergoing CT/CT angiography | 2 hours
  ct and ct angiography for exclusion of any bleeding or head injury

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wahlgren N, Ahmed N, Davalos A, Ford GA, Grond M, Hacke W, Hennerici MG, Kaste M, Kuelkens S, Larrue V, Lees KR, Roine RO, Soinne L, Toni D, Vanhooren G; SITS-MOST investigators. Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet. 2007 Jan 27;369(9558):275-82. doi: 10.1016/S0140-6736(07)60149-4. PMID 17258667